CLINICAL TRIAL: NCT03039712
Title: Longitudinal Coverage With Evidence Development Study on Micra Leadless Pacemakers
Acronym: Micra CED
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Micra CED Study
Record Dates: First submitted 2017-01-27; First posted 2017-02-01 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Micra leadless pacemaker therapy: All Medicare patients implanted with Micra leadless pacemaker system
- Single Chamber Transvenous pacemaker: All Medicare patients implanted with full system (e.g. lead and generator) single- chamber ventricular transvenous pacemakers

SUMMARY:
The primary purpose of the study is to meet the CMS mandated Coverage with Evidence Development requirement in the National Coverage Determination for Leadless Pacemakers as they apply to Medtronic Micra devices. The study uses administrative claims data of the Medicare population implanted with single-chamber ventricular pacemakers. Patients are enrolled through submission of claims or encounter data to CMS.

DETAILED DESCRIPTION:
Micra CED study is a study of the Medicare beneficiary population implanted with single-chamber ventricular pacemakers, and will be executed by analyzing administrative claims data. The study consists of two primary objectives: estimate the: (1) acute overall complication rate and (2) the 2-year survival rate of patients implanted with a Micra leadless pacemaker. As part of the secondary objectives of the study, a comparative analysis of Micra leadless pacemakers to single-chamber ventricular transvenous pacemakers will be conducted.

The analysis will be in CMS claims data and is subject to a central IRB. However, individual hospitals are not engaged in research and local IRB oversight is not necessary.

ELIGIBILITY:
Inclusion Criteria:

• Medicare beneficiaries implanted with a leadless pacemaker (CPT 0387T or 33274 or ICD-10 PCS 02HK3NZ) on or after the study start date will be included in the study.

or

• Medicare beneficiaries with implanted with a full system single-chamber ventricular transvenous pacemaker (CPT 33207 or ICD-10 PCS 0JH605Z or 0JH604Z and 02HK3JZ) on or after the study start date.

Exclusion Criteria:

• None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study cohort will include all Medicare patients with continuous claims data implanted with a Micra leadless pacemaker or a full-system single-chamber ventricular transvenous pacemaker in any US location.
Sampling Method: Probability Sample
Enrollment: 37000 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Acute complication rate | 30 days
  Single-chamber ventricular pacemaker system and/or procedure related complications at 30 days. Acute complications include embolism/thrombosis, event at the puncture site, cardiac effusion/perforation, device-related complication, or other complications following the implantation of a single-chamber ventricular pacemaker system. Subjects' administrative claims data will be reviewed to determine the occurrence of an acute complication.
The 2-year survival rate of patients implanted with a Micra leadless pacemaker | 2 years
  Estimate the 2-year survival rate of patients implanted with a Micra leadless pacemaker

SECONDARY OUTCOMES:
Chronic complication rate | 6 months
  Chronic complications are a subset of acute complications that may also occur within six months following the implantation of a single-chamber ventricular pacemaker. Single-chamber ventricular pacemaker system and/or procedure related complications at six months. Subjects' administrative claims data will be reviewed to determine the occurrence of a chronic complication.
Device-related re-intervention rates | 2 years
  Device-related re-interventions are procedures associated with the insertion/replacement, revision, or removal of either a leadless or transvenous pacemaker system or components following the index implantation of a single-chamber ventricular pacemaker. Device-related re-intervention rates will be reported at six month intervals for two years following the index implantation of a single-chamber ventricular pacemaker. Subjects' administrative claims data will be reviewed to determine the occurrence of a device-related re-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mikhael El Chami, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crossley GH, Piccini JP, Longacre C, Higuera L, Stromberg K, El-Chami MF. Leadless versus transvenous single-chamber ventricular pacemakers: 3 year follow-up of the Micra CED study. J Cardiovasc Electrophysiol. 2023 Apr;34(4):1015-1023. doi: 10.1111/jce.15863. Epub 2023 Feb 23. PMID 36807378
- [Derived] Boveda S, Higuera L, Longacre C, Wolff C, Wherry K, Stromberg K, El-Chami MF. Two-year outcomes of leadless vs. transvenous single-chamber ventricular pacemaker in high-risk subgroups. Europace. 2023 Mar 30;25(3):1041-1050. doi: 10.1093/europace/euad016. PMID 36757859
- [Derived] El-Chami MF, Bockstedt L, Longacre C, Higuera L, Stromberg K, Crossley G, Kowal RC, Piccini JP. Leadless vs. transvenous single-chamber ventricular pacing in the Micra CED study: 2-year follow-up. Eur Heart J. 2022 Mar 21;43(12):1207-1215. doi: 10.1093/eurheartj/ehab767. PMID 34788416